CLINICAL TRIAL: NCT07278713
Title: Effect of an Internet-Based, Mobile Terminal-Supported, Family-Participatory Early Rehabilitation Model on Sleep Improvement and Stigma Prevention in Critically Ill Patients: A Randomized Controlled Trial
Brief Title: Family-Participatory Early Rehabilitation in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qiao Ke, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022S00433
Record Dates: First submitted 2025-11-18; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Based, Family-Participatory Early Rehabilitation (IFPER) Group (Experimental): In addition to standard care, patients received a structured, family-participatory early rehabilitation program guided by the "7P Rehabilitation Pyramid Model." Trained family members used a mobile application to assist with activities including Position Management, Pain & Sedation Management, Physiotherapeutics, Pulmonary Rehabilitation, Psychological Rehabilitation, Performance Rebuilding, and fostering Purpose & Belonging. The sessions were conducted for 30-45 minutes, twice daily.
  Interventions: Behavioral: Internet-Based, Family-Participatory Early Rehabilitation (IFPER)
- Standard Care Group (Active Comparator): Patients received routine ICU care, which included standard medical and supportive care, daily assessments, sedation management, pain control, nutritional support, and standard early rehabilitation protocols delivered by the ICU physical therapy team.
  Interventions: Behavioral: Standard ICU Care

INTERVENTIONS:
Behavioral: Internet-Based, Family-Participatory Early Rehabilitation (IFPER) — A structured, multi-component rehabilitation program facilitated by trained family members using a mobile application for guidance and communication, based on the "7P Rehabilitation Model."
  Arms: Internet-Based, Family-Participatory Early Rehabilitation (IFPER) Group
Behavioral: Standard ICU Care — Routine ICU care including medical support and standard rehabilitation delivered by ICU staff.
  Arms: Standard Care Group

SUMMARY:
This prospective, randomized controlled trial aims to evaluate the efficacy of an Internet-Based, Family-Participatory Early Rehabilitation (IFPER) model compared to standard care for critically ill patients in the Intensive Care Unit (ICU). The study will determine if the IFPER model, which is based on a structured "7P Rehabilitation" framework, can improve sleep quality, reduce the perception of critical illness-related social stigma, and alleviate procedural pain.

DETAILED DESCRIPTION:
Critically ill patients often suffer from Post-Intensive Care Syndrome (PICS), which includes severe sleep disturbances, pain, and psychological issues like social stigma. While family involvement in care is known to be beneficial, structured, technology-supported models are scarce. This study was designed to address this gap by testing a novel IFPER model. A total of 204 adult patients admitted to the ICU were randomized to either the IFPER group or a standard care group. The IFPER intervention involves trained family members using a mobile application to deliver a structured, multi-component rehabilitation program based on the "7P Rehabilitation Model" (Position Management, Pain & Sedation, Physiotherapeutics, Pulmonary Rehabilitation, Psychological Rehabilitation, Performance Rebuilding, Purpose & Belonging). The standard care group received routine ICU care. The study hypothesizes that this structured, family-centered approach will lead to significantly better outcomes in sleep, stigma perception, and pain management compared to standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Expected ICU stay of more than 48 hours
* Hemodynamic stability (mean arterial pressure 65-110 mmHg with no or low-dose vasopressor support)
* Stable respiratory status (PaO2/FiO2 > 200 mmHg, SpO2 ≥ 88%)
* Richmond Agitation-Sedation Scale (RASS) score ≥ -2
* Having at least one family member willing and able to participate

Exclusion Criteria:

* Unstable cardiovascular conditions (e.g., acute coronary syndrome, malignant arrhythmia)
* Acute neurological injury with unstable intracranial pressure
* Unstable fractures or spinal cord injury
* Active, uncontrolled bleeding
* Pre-existing severe psychiatric disorders or dementia
* Inability to provide consent and no available legal surrogate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Sleep Efficiency | From enrollment through ICU discharge, an average of 10 days
  Measured by polysomnography (PSG). Sleep efficiency is calculated as (total sleep time / time in bed) × 100%. The change is assessed from baseline to the day before ICU discharge.

SECONDARY OUTCOMES:
Social Stigma Score | At ICU discharge, an average of 10 days after enrollment
  Measured by the Social Stigma in Critical Illness (SSCI) scale. The scale ranges from 10 to 50. A higher score indicates a worse outcome (greater perceived stigma).
Procedural Pain Scores | Through ICU stay, an average of 10 days
  Assessed daily using the Numeric Rating Scale (NRS) for communicative patients and the Critical-Care Pain Observation Tool (CPOT) for non-communicative patients. The NRS is on a 0-10 scale, and the CPOT is on a 0-8 scale. For both scales, a higher score indicates a worse outcome (more pain).
Duration of Mechanical Ventilation | Through ICU stay, an average of 7 days
  The total number of days a patient requires mechanical ventilation.
ICU Length of Stay | Through study completion, an average of 10 days
  The total number of days a patient stays in the ICU.
Incidence of Delirium | Through ICU stay, an average of 10 days
  The percentage of patients who develop delirium, assessed twice daily using the Confusion Assessment Method for the ICU (CAM-ICU).
Change in Percentage of REM Sleep | From enrollment through ICU discharge, an average of 10 days
  Change in the percentage of Rapid Eye Movement (REM) sleep, measured by polysomnography (PSG).
Change in Percentage of N1 Sleep | From enrollment through ICU discharge, an average of 10 days
  Change in the percentage of Stage 1 non-REM sleep, measured by polysomnography (PSG).
Change in Percentage of N2 Sleep | From enrollment through ICU discharge, an average of 10 days
  Change in the percentage of Stage 3 non-REM (slow-wave) sleep, measured by polysomnography (PSG).
Change in Arousal Index | From enrollment through ICU discharge, an average of 10 days
  Change in the number of arousals or awakenings per hour of sleep, measured by polysomnography (PSG).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China